CLINICAL TRIAL: NCT06628843
Title: Twin Vaginal Deliveries and Maternal-fetal Outcomes Before and After Starting Training of Teamworks
Brief Title: Twin Vaginal Breech Deliveries Before and After Starting Training Skills and Clinical Approach in Labor Ward
Acronym: TVBD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: G. d'Annunzio University (Other)
Collaborators: San Giovanni di Dio Hospital (Other)
Responsible Party: Principal Investigator, Claudio Celentano, MD, G. d'Annunzio University
Other Study IDs: ObGynEASC007
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-01

CONDITIONS: Cearean Section Rate; Maternal Adverse Outcomes; Neonatal Adverse Outcomes
Keywords: Twin vaginal birth; PPH; NICU stay

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Before: twin deliveries after 34 wks 2017 january-2020 December (Pescara), and 2020 January-2022 June (Florence)
  Interventions: Other: cesarean section rate
- After: twin deliveries after 34 wks January 2021-december 2024 (Pescara), and July 2022-December 2024
  Interventions: Other: cesarean section rate

INTERVENTIONS:
Other: cesarean section rate — Incidence of cesarean sections in the two periods, Rate of adverse outcomes within vaginal and cesarean deliveries

SUMMARY:
In January 2021 Dept of ObGyn of Santo Spirito Hospital Pescara Italy, and in July 2022 Dept of ObGyn of San Giovanni di Dio Hospital Florence Italy, started regular training in management of obstetric emergencies. Twin vaginal deliveries were considered when first fetus is vertex presenting. The present study is evaluating retrospectively the rate of vaginal birth in twins after 34 weeks' gestation in the period 2017-2020, and 2021-2024 for Santo Spirito Hospital Pescara, and 2020-2022 June, and July 2022-2024 for San Giovanni di Dio Hospital Pescara. Incidence of maternal and fetal/neonatal outcomes were considered. Policy in Pescara hospital is based on cultural support of teamworks working in labor ward. Florence policy is based on availability of two teamworks previously skilled for twin vaginal delivery

DETAILED DESCRIPTION:
In the period 2017-2020 before starting of simulator training for obstetrics emergencies, twin birth were collected. Incidence of vaginal birth and incidence of maternal adverse outcome (such as PPH) and fetal/neonatal adverse outcome (such as NICU stay) were recorded. The same outcomes were collected in twin deliveries after 34 wks in the period 2021-2024. Similarly in San Giovanni di Dio Hospital Florence they started this protocol in July 2022. The retrospective data enrollement identified the period January 2020-June 2022 and July 2022-December 2024. Teamworks in Pescara Hospital were supported by continous formation for retaining skills on vaginal birth particularly twin vaginal deliveries. In Florence Hospital two teamworks were supporting patients wondering for a vaginal birth and in the meantime positive results were collected in labor ward

ELIGIBILITY:
Inclusion Criteria:

* twin pregnancies after 34 weeks

Exclusion Criteria:

* multiple pregnancies monochorionic monoamniotic pregnancies gestational age before 34 weeks completed cesarean indication unrelated to pregnancy (placenta previa, maternal diseases, etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with twin pregnancies after 34 weeks' gestation
Study Population: Pregnancies after 34 weeks' gestation elegible for vaginal birth
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal birth | 4 years (Pescara)- 2.5 years (Florence)
  Rate of vaginal birth

SECONDARY OUTCOMES:
Maternal outcomes | 4 years (Pescara)- 2.5 years (Florence)
  Rate of PPH within cesarean section and vaginal deliveries
Fetal Neonatal outcomes | 4 years (Pescara)- 2.5 years (Florence)
  Incidence of overall fetal neonatal outcomes (such as NICU stay, RDS, HPE, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Celentano, MD, Principal Investigator — University d'Annunzio Chieti Pescara
Locations (2):
- Italy (2):
  - San Giovanni di Dio Hospital, Florence, FI
  - Santo Spirito Hospital, Pescara, PE

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: University website — http://www.unich.it